CLINICAL TRIAL: NCT07204717
Title: Ring Free Gingival Techniqea :A Randomized Controlled Trial
Brief Title: Ring Free Gingival Techniqea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra ATEŞ (Other)
Responsible Party: Sponsor-Investigator, Esra ATEŞ, assistant professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Abant IBU.
Record Dates: First submitted 2025-09-19; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Free Gingival Graft Volume Change
Keywords: Dental Implant; Keratinized Mucosa.; Rıng free gingival graft; Free gingival graft

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ring free gingival graft (Experimental): ring free gingival graft
  Interventions: Procedure: ring free gingival greft
- standard free gingival technique (Active Comparator): standard techinique
  Interventions: Procedure: free gingival graft

INTERVENTIONS:
Procedure: free gingival graft — standard free gingival technique
  Arms: standard free gingival technique
Procedure: ring free gingival greft — ring free gingival greft technique
  Other Names: ring free gingival
  Arms: ring free gingival graft

SUMMARY:
Objective Peri-implant keratinized mucosa deficiency is a significant factor affecting implant success. Therefore, it is crucial to choose a suitable technique for increasing the width of the keratinized mucosa. This study aims to compare two different approaches of free gingival graft (FGG) application in the treatment of insufficient peri-implant keratinized mucosa and to determine the most effective and predictable technique.

Materials and Methods A total of 38 systemically healthy patients with ≤2 mm of keratinized mucosa in the mandibular anterior region (teeth 33-43) and 38 dental implants were included. Patients were randomly assigned to two groups: Test ( Ring FGG) and Control (Conventional FGG). Clinical parameters including Bleeding on Probing (BOP), Gingival Index (GI), Plaque Index (PI), Probing Depth (PD), Width of Keratinized Mucosa (KMW), Peri-implant Mucosal Thickness (PMT), and Graft Surface Area (GSA) were recorded at baseline, and at 1, 3, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 1. Systemically healthy individuals 2. Age over 18 years 3. Non-smokers 4. No antibiotic therapy for any reason in the past 6 months 5. No previous soft tissue surgery performed in the region of interest 6. KMW≤ 2 mm 7. Presence of inadequate keratinized tissue in the vestibular and/or lingual area of the anterior mandibular implant region 8. Mentally competent to understand the study purpose and procedures explained both verbally and in writing

Exclusion Criteria:

- 1. Presence of peri-implantitis in the implant(s) planned for FGG application (defined as probing depth ≥ 5 mm, pus discharge, mobility, or severe bone loss) 2. Inability to maintain oral hygiene or presence of implant body and/or abutment fractures in the related region 3. Presence of pathological conditions in the palate that prevent harvesting of a free gingival graft 4. History of systemic diseases such as Diabetes Mellitus, Chronic Renal Failure, Cancer, Bleeding Disorders, Connective Tissue Diseases, etc.

5. Use of anticoagulant and/or antiplatelet medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 38 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
keratinize gingiva | 2 week
  increasing the amount of keratinized gingiva

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Bolu Abant İzzet Baysal University,, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP